CLINICAL TRIAL: NCT05858710
Title: Phase I Dose Escalation Study of 3-Weekly Intravenous DPPG2-TSL-DOX Combined With Regional Hyperthermia in Locally Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Study of DPPG2-TSL-DOX Combined With Hyperthermia in Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thermosome GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS-DM-STS-101; 2023-507836-19-00 (EU CTIS Number); 2020-005033-32 (EudraCT Number)
Record Dates: First submitted 2023-04-24; First posted 2023-05-15 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue; Doxorubicin/ IV + Liposomes; Doxorubicin
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Dexrazoxane

STUDY DESIGN:
Intervention Model Description: an adapted 3+3 multiple ascending dose (MAD) design with sentinel dosing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV DPPG2-TSL-DOX (Experimental): DPPG2-TSL-DOX (20 or 40 or 50 mg/m^2) + regional hyperthermia (RHT)
  3 dose levels are planned in this study: dose level 1 will be receiving 20 mg/m^2 DPPG2-TSL-DOX, dose level 2 will be receiving 40 mg/m^2 DPPG2-TSL-DOX, dose level 3 will be receiving 50 mg/m^2 DPPG2-TSL-DOX.
  Participants are to be treated with DPPG2-TSL-DOX infusion over 30 minutes and RHT every three weeks (one cycle = 21 days), receiving up to 6 cycles in Main Study Phase and additional 6 cycles in Treatment Continuation Phase, if eligible:
  * In the first cycle (cycle 1), DPPG2-TSL-DOX application will be performed without RHT in all participants for safety precaution.
  * In cycles 2-12, DPPG2-TSL-DOX will be applied in parallel with RHT. Dexrazoxane as cardioprotectant will be provided for participants overcoming a cumulative dose of 300 mg/m^2 DOX.
  Interventions: Drug: DPPG2-TSL-DOX; Drug: Dexrazoxane

INTERVENTIONS:
Drug: DPPG2-TSL-DOX — DPPG2-TSL-DOX is a thermosensitive liposomal formulation of doxorubicin.
  Other Names: Doxorubicin; THE001
Drug: Dexrazoxane — For cardioprotection of participants.

SUMMARY:
This study aims to explore a new therapeutic approach for advanced soft tissue sarcoma (STS) by investigating the safety, tolerability, and maximum tolerated dose (MTD)/highest tolerated dose (HTD) of DPPG2-TSL-DOX combined with regional hyperthermia (RHT) in patients who have been pre-treated with anthracycline, e.g. doxorubicin (DOX).

DETAILED DESCRIPTION:
Considering that up to 40 percentage of patients with soft tissue sarcoma (STS) will develop metastatic disease and that for these patients overall survival (OS) ranges between 3.7 to 25 months it becomes clear that new therapeutic approaches for the treatment of advanced STS are urgently needed. Doxorubicin (DOX) is a cytotoxic compound that belongs to the class of anthracyclines. DOX has had market authorization since 1960s and is considered the most active chemotherapeutic drug for the treatment of STS. DPPG2-TSL-DOX is a novel formulation of DOX encapsulated in DPPG2-containing thermosensitive liposomes (TSL). Regional hyperthermia (RHT) with a tumor target temperature of ≥41.5 to ≤44 degree of Celsius combined with anthracycline-based chemotherapy has shown to improve survival in patients with localized high-risk STS. Treatment with DPPG2-TSL-DOX aims at combining the confirmed anti-tumor efficacy of anthracyclines in the treatment of locally advanced STS with RHT-triggered DOX release from circulating liposomes resulting in higher local DOX concentrations in the tumor as observed in preclinical studies.

DPPG2-TSL-DOX combined with RHT has been investigated in feline sarcoma at 1 mg/kg dose level resembling the clinically recommended dose level of standard DOX with considerably improved efficacy and better tolerability. The proposed study will characterize the safety and tolerability and, if applicable, the maximum tolerated dose (MTD)/highest tolerated dose (HTD) of DPPG2-TSL-DOX in combination with RHT in patients with advanced or metastatic STS who have been pre-treated with anthracycline. An adapted 3+3 MAD study design with sentinel dosing and a starting dose of 20 mg/m^2 DPPG2-TSL-DOX is applied in this study to identify dose-limiting toxicities (DLTs) of DPPG2-TSL-DOX in combination with RHT.

ELIGIBILITY:
Inclusion criteria

1. Age at the time of consent ≥18 years.
2. Patient has provided written informed consent prior to any study-specific procedure.
3. Locally advanced (unresectable) or metastatic STS, including histological sarcoma subtypes treated as STS, for which treatment with DOX monotherapy is appropriate, as confirmed by the investigator.
4. Pretreatment with an anthracycline (including DOX, epirubicin as mono- or combination therapy). Patients who received anthracycline in an adjuvant setting are eligible.
5. Progressive disease not suitable for surgery after

   1. only one further line of chemotherapy (including TKI) if the RHT field targets the clinically relevant tumor manifestation/s (e.g., locally advanced or multifocal intraabdominal STS; diffuse metastatic STS in which RHT of a tumor manifestation [e.g., liver] is considered relevant although other systemic metastases are present that do not endanger the patient, as per the judgment of the investigator), or
   2. two or more further lines of chemotherapies (including TKI) for patients with metastatic STS and a tumor manifestation suitable for RHT.
6. All previous oncological treatments must have been completed ≥3 weeks (21 days) prior to the first dose of study treatment, ensuring a sufficient washout period.
7. Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (Eisenhauer et al. 2009).
8. Tumor accessible for RHT.
9. Left ventricular ejection fraction (LVEF) >50% (within 28 days prior to enrolment).
10. Adequate hematologic, organ and coagulation function within 14 days prior to enrolment as assessed by local lab:

    1. Absolute neutrophil count (ANC) ≥1.5×10^9/L. Granulocyte-colony stimulating factor (G-CSF) cannot be administered within 2 weeks (14 days) prior to enrolment.
    2. Platelet count ≥100×10^9/L.
    3. Hemoglobin ≥9.0 g/dL. No transfusions are allowed within 2 weeks (14 days) prior to enrolment.
    4. Serum creatinine ≤1.5 times upper limit of normal (ULN).
    5. Negative dipstick for proteinuria or if proteinuria ≥2+ (equals ≥ 1001 mg/L or 1.001 g/L (Lamb, et al., 2009), then additional 24 h urine collection <1g protein/ 24 h.
    6. Total bilirubin within ULN (except for patients with Gilbert's syndrome, who must have a total bilirubin <3 mg/dL).
    7. ALT/ AST ≤3.0×ULN; if the liver has tumor involvement, AST and ALT ≤5.0×ULN are acceptable.
    8. An adequate coagulation function as defined by international normalized ratio (INR) ≤1.5×ULN or prothrombin time ≤1.5×ULN, and partial thromboplastin time ≤1.5×ULN (unless receiving anticoagulant therapy). Patients receiving phenprocoumon are recommended to switch to low molecular weight heparin and should have achieved stable coagulation status prior to the first dose of study treatment.
11. Tubular excretion rate (TER) by MAG-3-clearance ≥ TERLoLi (TERLoLi = 70% TERNorm).
12. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (Appendix 1).
13. If female, must:

    1. Be not of child-bearing potential due to surgical sterilization (at least 6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history or menopause.
    2. Be a post-menopausal woman, defined as a woman meeting either of the following criteria:

    i. spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (for example, oral contraceptives, hormones, gonadotropin-releasing hormone, antiestrogens, selective estrogen receptor modulators [SERMs], or chemotherapy) ii. spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone level >40 mIU/mL.
14. Women of childbearing potential (WOCBP; for a definition see Appendix 2) and men able to father a child must be ready and able to use two medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at screening, during trial participation, and until 6 months after last dose of study treatment. Also, partner of male participants, who is of childbearing potential must use a highly effective method of contraception during the same duration (Please refer to Appendix 2 for methods of highly effective contraception). A list of contraception methods meeting these criteria is provided in the patient information.
15. At least 3 months' life expectancy in the investigator's assessment.

Exclusion criteria

1. Patients already enrolled in any clinical study involving an investigational product or medical device or have participated within the past 30 days in a clinical trial involving an investigational product or medical device.
2. History of another primary malignancy, with the exception of:

   1. curatively treated non-melanomatous skin cancer
   2. curatively treated cervical carcinoma in situ
   3. non-metastatic prostate cancer, or
   4. other primary non-hematologic malignancies that had been treated with curative intent, no known active disease, and no treatment administered during the last 3 years prior to enrolment that the investigator agrees will not affect the interpretation of study results or would be unsuitable for participation in the study.
3. Active fungal, bacterial and/or known viral infection including human immunodeficiency virus or viral (A, B, or C) hepatitis.
4. Resting heart rate of >100 bpm (measured after ≥10 min. in seated position). Note: If >100 bpm, the measurement should be repeated by up to 3 consecutive measurements at least 10 minutes apart from each other. If all 3 measurements are >100 bpm the exclusion criterion is met.
5. Uncontrolled intercurrent illness including, but not limited to, an ongoing/active infection requiring parenteral antibiotics.
6. Have a serious cardiac condition, such as:

   1. unstable angina pectoris
   2. angioplasty, cardiac stenting, or myocardial infarction within 6 months of enrolment
   3. valvulopathy that is severe, moderate, or deemed clinically significant
   4. arrhythmias that are symptomatic or require treatment
7. Have a QTcF interval of >450 msec for males and >470 msec for females on screening electrocardiogram (ECG) utilizing Fridericia's correction.
8. Psychiatric illness or social situation that would limit compliance with study requirements.
9. Any planned or required major surgery during the course of the study.
10. Pregnant or breastfeeding female.
11. Individuals who are institutionalized on a judicial or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | End of study (up to 14 months)
  If no more than 1 subject experiencing DLTs is identified after all subjects completed cycle 3 in dose level 3, MTD for the current study and study population will be considered 50 mg/m2.
Highest tolerated dose (HTD) | End of study (up to 14 months)
  Highest dose considered safe for dose escalation by the independent DSMB in the FiH study provided < 33% experiencing a DLT per DL are reported in the study until completion or early termination.

SECONDARY OUTCOMES:
Adverse Events (AEs) | End of study (up to 14 months)
  Number of treatment-emergent AEs according to CTCAE 5.0
Serious Adverse Events (SAEs) | End of study (up to 14 months)
  Number of treatment-emergent SAEs according to CTCAE 5.0
Laboratory abnormalities | End of study (up to 14 months)
  Number of laboratory abnormalities
Electrocardiogram (ECG) abnormalities | End of study (up to 14 months)
  Number of participants with ECG abnormalities
Echocardiogram (ECHO) abnormalities | End of study (up to 14 months)
  Number of participants with ECHO abnormalities
Renal toxicities | End of study (up to 14 months)
  Number of participants with renal toxicities
Maximum concentration (Cmax) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Last measurable (non-zero) concentration (Clast) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Area under the curve from time 0 to x hours (AUC[0-x] ) after the start of infusion of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Area under the curve from time 0 to the time of the last quantifiable concentration (AUC[0-tlast) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Time of maximum observed concentration (Tmax) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Terminal half-life (T½) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Clearance (CL) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Volume of distribution at steady-state (Vss) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  without RHT (cycle 1; 12 time points)
Maximum concentration obtained after administration (Cmax) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Last measurable (non-zero) concentration (Clast) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Area under the curve from time 0 to x hours (AUC[0-x] ) after the start of infusion of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Area under the curve from time 0 to the time of the last quantifiable concentration (AUC[0-tlast) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Time of maximum observed concentration (Tmax) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Terminal half-life (T½) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Clearance (CL) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)
Volume of distribution at steady-state (Vss) of DPPG2, non-liposomal DOX, liposomal encapsulated DOX and total DOX | End of study (upto 14 months)
  with RHT (cycle 2; 12 time points)

OTHER OUTCOMES:
Radiographic response | day 64 (+/-3) in the study for each participant and end of study (21 [+7] days after last study drug treatment)
  Radiographic response rates (CR, PR, SD, PD) and ORR (CR+PR) as assessed by RECIST 1.1
Radiographic local response | day 64 (+/-3) in the study for each participant and end of study (21 [+7] days after last study drug treatment)
  Radiographic local response rates (CR, PR, SD, PD) by Choi et al. 2007 assessed for target and non-target lesions in RHT field
Tumor temperatures (optional) | day 23, 44, 65, 86, 107 (+/-3) in the study for each participant
  Specific tumor temperature parameters: Tmax, T90, T50, T20 and respective cumulative minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reichardt, PD Dr., Principal Investigator — Helios Klinikum Berlin-Buch GmbH
Locations (2):
- Germany (2):
  - Helios Klinikum Berlin-Buch GmbH, Berlin
  - Klinikum der Universität München (KUM) Campus Großhadern, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website giving information on the drug technology — https://www.thermosome.com/